CLINICAL TRIAL: NCT06794437
Title: Turkish Version of Mobile Device Proficiency Questionnaire, Validity and Reliability Study
Brief Title: Turkish Version of Mobile Device Proficiency Questionnaire
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Principal Investigator, Uludag University
Other Study IDs: 2025/1-4
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Geriatric; Technology
Keywords: MDPQ; Reliability; Validity; MDPQ-TR
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Translate and culturally adapt the original English version of the Mobile Device Proficiency Questionnaire

SUMMARY:
The Mobile Device Proficiency Questionnaire (MDPQ) contains 46 questions with eight subscales, which are as follows: mobile device basics, communication, data and file storage, internet, calendar, entertainment, privacy, and troubleshooting and software management. Each question item is rated on a five-point scale based on the individual's subjective proficiency level. The scores ranged from 8 to 40 and were scored in a similar manner to in the original version. For each subscale of the MDPQ, responses for all questions were averaged. These averaged scores were then summed across subscales to come up with a total score of the MDPQ.

DETAILED DESCRIPTION:
Information and Communication Technologies (ICT) enable users to perform various tasks with minimal effort. Today, many elderly individuals also own their own mobile devices. Mobile devices are small, lightweight and portable information terminals, and are indispensable for ICT use in our daily lives with models such as smartphones and tablet computers. In addition, in the USA and Japan, 61% and 74.2% of individuals aged 65 and over use smartphones, respectively. Mobile devices are used for various functions in daily life such as making phone calls, messaging, checking programs, shopping, paying bills and accessing entertainment content, facilitating many tasks. However, some elderly individuals who own mobile devices do not sufficiently benefit from the advantages offered by ICT. There are significant differences in internet literacy among elderly individuals, and social and socioeconomic factors can affect the digital gap among elderly individuals. Due to these social factors, efforts to eliminate digital inequality need to be increased in the future.

This study aims to adapt the Mobile Device Proficiency Questionnaires (MDPQ) to Turkish. MDPQ can serve as a basic and quantitative indicator of ICT proficiency among the elderly population. In this context, the Turkish version of MDPQ, MDPQ-T, will be created and its reliability and validity will be verified. We expect this new assessment tool to have the same high reliability and validity as the original version in the Turkish population. We also predict that the duration or frequency of use of mobile devices will be positively correlated with mobile device proficiency measured by MDPQ-T. In addition, we expect not only the accessibility of mobile devices but also the subjective importance, performance and satisfaction level of mobile device use in daily life to be positively correlated with MDPQ-T.

ELIGIBILITY:
Inclusion Criteria:

* Being a native Turkish speaker,
* Having no reading or writing problems,
* Having a mobile device such as a phone or tablet,
* Agreeing to participate in the study

Exclusion Criteria:

* Individuals with neurological diseases such as cognitive impairment, Alzheimer's, dementia, etc. will be excluded from the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Geriatric individuals between the ages of 65-80
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Age of the patients | 1 week
  Age will be recorded.
Gender of the patients | 1 week
  Gender will be recorded.
education level of the patients | 1 week
  education level will be recorded
Mobile Device Proficiency Questionnaire | 1 week
  Mobile Device Proficiency Questionnaire will be filled out under the supervision of a physiotherapist
system usability scale Questionnaire | 1 week
  system usability scale Questionnaire will be filled out under the supervision of a physiotherapist

CONTACTS AND LOCATIONS:
Overall Officials: Selim Mahmut GÜNAY, Dr, Study Chair — Uludağ University
Locations (1):
- Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided